CLINICAL TRIAL: NCT05583591
Title: Prospective, Randomized Controlled Study Comparing Combined Phacoemulsification With iStent Inject W Versus Hydrus for Mild to Moderate Open Angle Glaucoma (COMPETE)
Brief Title: Combined Phacoemulsification With iStent Inject W Versus Hydrus for Mild to Moderate Open Angle Glaucoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment, sites unable to obtain iStent Inject W from manufacturer
Sponsor: Diablo Eye Associates (Industry)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COMPETE Trial
Record Dates: First submitted 2022-10-14; First posted 2022-10-17 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Open Angle Glaucoma
Keywords: Primary Open Angle Glaucoma; Hydrus; iStent; minimally invasive glaucoma surgery; MIGS; randomized
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Combined cataract surgery with Hydrus microstent (Active Comparator)
  Interventions: Device: Combined cataract surgery with Hydrus microstent; Device: Combined cataract surgery with iStent Inject W
- Combined cataract surgery with iStent Inject W (Active Comparator)
  Interventions: Device: Combined cataract surgery with Hydrus microstent; Device: Combined cataract surgery with iStent Inject W

INTERVENTIONS:
Device: Combined cataract surgery with Hydrus microstent — Device designed to help lower intraocular pressure by improving aqueous outflow through the trabecular meshwork. Used in combination with cataract surgery.
Device: Combined cataract surgery with iStent Inject W — Device designed to help lower intraocular pressure by improving aqueous outflow through the trabecular meshwork. Used in combination with cataract surgery.

SUMMARY:
The goal of the study is to prospectively evaluate and compare Hydrus microstent to the iStent Inject Wide in combination with cataract surgery in patients with mild to moderate open angle glaucoma. Hydrus and iStent are the two FDA approved trabecular meshwork targeting microstents to treat open angle glaucoma in conjunction with cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* >60 years or older
* Visually significant cataract
* Mild to moderate primary open angle glaucoma controlled on medications
* undergoing cataract surgery with lens implantation and concurrent microstent placement
* IOP ≥ 21 mmHg and ≤ 36 mmHg after washout of ocular hypotensive medication(s)
* CCT 480 to 620μm
* No prior ocular surgery including corneal refractive surgery
* No SLT within 6 months of baseline visit, no history of intracameral glaucoma drug eluting implants
* Visual field mean deviation ≤ -12 dB
* Optic nerve abnormalities consistent with glaucoma, C/D ratio less than ≤0.8

Exclusion Criteria:

* Prior intraocular surgery
* Visual field MD ≥ -12 dB
* secondary glaucoma including uveitis, traumatic, malignant, neovascular, and congenital glaucoma.
* Glaucoma related to elevated episcleral venous pressure including Sturge-Weber syndrome, thyroid eye disease, orbital tumor, and etc.
* Uncontrolled intraocular pressure on maximum tolerated medical therapy;
* Unable to perform wash-out IOP
* Anatomic exclusion of narrow anterior chamber angle (Shaffer grade I-II), other angle abnormalities including angle closure glaucoma
* Corneal disease or dystrophy
* Pathological myopia with degeneration that affects diagnostic imaging
* Clinically significant ocular pathology or degenerative diseases that affect vision, visual field, or optical coherence tomography of optic nerve.
* Inability to perform reliable Visual Field and optical coherence tomography.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with complete success defined as intraocular pressure reduction > 25% from baseline And without secondary intervention to reduce IOP (medication, laser trabeculoplasty, or surgery) at 24 month. | 24 Months

SECONDARY OUTCOMES:
Intraoperative and postoperative adverse events rates | 24 Months
Rates of secondary intervention to reduce intraocular pressure | 24 Months
Rates of needing incisional glaucoma surgery as secondary intervention to control interocular pressure | 24 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Diablo Eye Associates, Walnut Creek, California, United States